CLINICAL TRIAL: NCT02773667
Title: Relationship Between Estimated Glomerular Filtration Rate and Biological Half-life of 131I. Prospective Analysis in Patients With Differentiated Thyroid Carcinoma.
Brief Title: Renal Tracer Elimination in Thyroid Cancer Patients Treated With 131-Iodine
Acronym: RETENTION
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: I-131-07/2015
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Correlation analysis between estimated renal function and biological half life of 131-I during radioiodine treatment of patients with differentiated thyroid cancer.

DETAILED DESCRIPTION:
131-I during radioiodine treatment of patients with differentiated thyroid cancer is mainly renally excreted. It is advised in the clinical guidelines that serum creatinine should be determined before applying 131-I and if necessary the administered dose should be reduced. Nevertheless no guideline gives advice in what extent the dose should be decreased. The adjustment is at the discretion of the attending physician.

Aim of this prospective study is to correlate the biological half life of 131-I with the renal function to give objective recommendations concerning the reduction of the applied dose in patients with limited renal function.

ELIGIBILITY:
Inclusion Criteria:

* patients with differentiated thyroid carcinoma
* stationary for treatment or diagnostic with radioiodine
* state after thyroidectomy
* written consent of the patient
* minimum age 18 years

Exclusion Criteria:

* no written consent of the patient
* patients with large residual thyroid tissue (iodine uptake > 10%)
* children under 18 years of age
* inclusion in concurrent interventional studies
* patients without TSH-stimulation by rhTSH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological secured differentiated thyroid cancer stationary for treatment or diagnostic with radioiodine
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-01; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Correlation between estimated renal function and biological half life of 131-I | 2 years
  The estimated renal function (estimated GFR) is measured via determination of serum creatinine and Cystatin C.
  The biological half-life of I-131 is determined via whole-body dosimetry (whole-body probe and whole-body gamma camera) and blood probe measurement.
  Update 2017/06/07: After analyzing the preliminary results (based on the first 48 patients) probe measurements are not longer needed in a simplified study design. Additionally, measuring the creatinine concentration is no longer needed in comparison to the Cystatin C measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Freesmeyer, Dr. med., Principal Investigator — Study Principal Investigator
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No